CLINICAL TRIAL: NCT03002675
Title: The Effect of Exenatide on Brown Adipose Tissue Activity and Energy Expenditure in Healthy Young Men
Brief Title: Exenatide and Brown Adipose Tissue
Acronym: exe01
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ingrid Jazet (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Ingrid Jazet, Dr, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P16.078
Record Dates: First submitted 2016-12-15; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: Adipose tissue; Type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exenatide (Experimental): Participants will receive exenatide (Bydureon, 2mg s.c. 1x/wk, AstraZeneca) during 12 weeks
  Interventions: Drug: Bydureon

INTERVENTIONS:
Drug: Bydureon — exenatide (Bydureon) 2mg s.c. 1x/wk
  Other Names: exenatide

SUMMARY:
The obesity epidemic has led to a enormous increase in the prevalence of type 2 diabetes mellitus (T2D), dyslipidemia and cardiovascular events. Particularly South Asians, who comprise 1/5 of the world population, are at increased risk of developing a disadvantageous metabolic phenotype and these diseases. Moreover, T2D occurs at a younger age and at a lower BMI when compared to white Caucasians. Recent research has shown that South Asians not only have a lower energy expenditure than their Caucasian counterparts, but also less active brown adipose tissue (BAT).

For some time, it has been known that adult humans have active BAT. This metabolic tissue produces heat by combusting triglycerides, in contrast to white adipose tissue, which stores this form of energy. It has been shown that activation of BAT has a positive effect on whole body metabolism, via increasing energy expenditure and improving glucose- and lipid metabolism. For this matter, BAT has been proposed as a major key player in energy homeostasis, which may be implemented in the current combat against the obesity epidemic. Aside from cold exposure, more research focuses on pharmacological activation of BAT.

Glucagon-like peptide 1 (GLP-1) is an incretin hormone which is produced by intestinal L-cells and upon food intake stimulates insulin secretion by pancreatic beta cells. The GLP-1 analogue Exenatide is a currently much used antidiabetic drug to reduce hyperglycemia via this aforementioned mechanism. Beyond its blood glucose-improving effects, Exenatide has also shown to lower body weight and improve dyslipidemia in T2D patients. Elucidation of the underlying mechanism of these beneficial effects is highly relevant.

Recent preclinical research in our group has shown that central activation of the GLP-1 receptor through exenatide increases BAT activity and thereby contributes to weight loss and improvement of dyslipidemia. The aim of this research project is to investigate whether exenatide is also able to activate BAT and increase resting energy expenditure, thereby improving glucose- and lipid metabolism and reducing fat mass and body weight in humans. Moreover, the investigators aim to validate the MRI scan as a novel way to measure BAT activity. The investigators hope that these forthcoming findings lead to the discovery of new treatment strategies against obesity.

DETAILED DESCRIPTION:
The current study is an open-label single arm prospective design, including 24 healthy young lean males (BMI between 18 and 25 kg/m2), of whom 12 Dutch South Asians and 12 Dutch Caucasians. After a medical screening, included subjects will receive 12 weeks of treatment with the GLP-1 analogue exenatide (Bydureon; 2 mg s.c. 1x/wk). Study subjects will visit the LUMC weekly. Before and after treatment there will be a study day, in which BAT (by means of 18F-FDG PET-CT scan and MRI scan), resting energy expenditure (measured by indirect calorimetry) and fat mass (by bio-impedance analysis) will be measured. Moreover, blood will be drawn to investigate the effects of exenatide on lipid- and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Dutch South Asian or white Caucasian male, 20-30 years
* BMI ≥ 18 and ≤ 25 kg/m2
* Good general health

Exclusion Criteria:

* BMI > 25 kg/m2 or < 18 kg/m2
* Use of medication known to influence glucose and/or lipid metabolism or brown fat activity (e.g. beta blockers)
* Any significant chronic disease
* Renal, hepatic or endocrine disease
* Smoking
* Participation in an intensive weight-loss program or vigorous exercise program during the last year before the start of the study
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year
* Contraindications for undergoing an MRI scan:
* Presence of non-MR safe metal implants or objects in the body.
* Pacemaker, neurostimulator, hydrocephalus pump, drug pump, non-removable hearing aid, large recent tattoos.
* Claustrophobia
* Tinnitus or hyperacusis

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The effect of exenatide on BAT activity and energy expenditure in healthy young South Asian compared to white Caucasian men | End of the study, up to 21 months

SECONDARY OUTCOMES:
Visualisation of BAT as measured with MRI scan compared to FDG-PET CT | End of the study, up to 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Jazet, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Janssen LGM, Nahon KJ, Bracke KFM, van den Broek D, Smit R, Sardjoe Mishre ASD, Koorneef LL, Martinez-Tellez B, Burakiewicz J, Kan HE, van Velden FHP, Pereira Arias-Bouda LM, de Geus-Oei LF, Berbee JFP, Jazet IM, Boon MR, Rensen PCN. Twelve weeks of exenatide treatment increases [18F]fluorodeoxyglucose uptake by brown adipose tissue without affecting oxidative resting energy expenditure in nondiabetic males. Metabolism. 2020 May;106:154167. doi: 10.1016/j.metabol.2020.154167. Epub 2020 Jan 23. PMID 31982480